CLINICAL TRIAL: NCT00555841
Title: Safety and Efficacy of Oral Acetyl-l-carnitine (ALC) in Non-anemic Potentially Curable Breast Cancer Subjects Undergoing Adjuvant Radiation Therapy Who Have Moderate to Severe Fatigue
Brief Title: Safety and Efficacy of ALC in Breast Cancer in Subjects With Fatigue
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: Sigma-Tau Research, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ST 03-103
Record Dates: First submitted 2007-11-07; First posted 2007-11-09 (Estimated); Last update posted 2012-08-28 (Estimated); Status verified 2012-08

CONDITIONS: Breast Cancer
Keywords: breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — allantoicase

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ALC (Experimental): I g three times daily
  Interventions: Drug: ALC and Placebo
- Placebo (Placebo Comparator): 1 g three times daily
  Interventions: Drug: ALC and Placebo

INTERVENTIONS:
Drug: ALC and Placebo — ALC and Placebo

SUMMARY:
The objective of this study is to evaluate the efficacy and safety of ALC in the treatment of non-anemic, breast cancer subjects who develop moderate or severe fatigue during adjuvant radiotherapy.

DETAILED DESCRIPTION:
The objective of this study is to evaluate the efficacy and safety of ALC in the treatment of non-anemic, breast cancer subjects who develop moderate or severe fatigue during adjuvant radiotherapy

ELIGIBILITY:
Inclusion Criteria:

* Stage 0-III breast cancer in which adjuvant radiation is indicated;
* Qualifying Brief Fatigue Inventory (BFI) score 6. -

Exclusion Criteria:

* Medication to treat or manage fatigue and pain
* Use of erythropoietin to control anemia
* Clinical evidence of hypothyroidism or hyperthyroidism

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2007-03; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
Change of BFI as evaluated from Baseline to Final Visit | 16 weeks

SECONDARY OUTCOMES:
Changes in Health-Related Quality of Life (HQoL) outcomes using Medical Outcomes Study Short Form Health Status Profile 12 items (MOS-SF 12 | 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Carmen Escalante, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- The University of Texas MD Anderson Cancer Center, Houston, Texas, United States